CLINICAL TRIAL: NCT03142321
Title: Defining Predictors of Radiological Transmural Response to Vedolizumab in Small Bowel Crohn's Disease Through Serum Proteomic Biomarkers
Brief Title: Defining Predictors of RT Response to Vedolizumab in IBD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201705043 -17-001
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease of Small Intestine
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vedolizumab 300 MG Injection [Entyvio] (Experimental): Vedolizumab will be initiated at 300 mg intravenous (IV) dosing at 0, 2 and 6 weeks followed by the 1st maintenance with 300 mg IV at week 14. Patients who have not achieved clinical response at week 14 will be eligible to undergo dose escalation to 4 weekly dosing of vedolizumab depending on the judgement of the treating gastroenterologist.
  Interventions: Drug: Vedolizumab 300 MG Injection [Entyvio]

INTERVENTIONS:
Drug: Vedolizumab 300 MG Injection [Entyvio] — Vedolizumab Injection
  Other Names: Entyvio

SUMMARY:
The overall goal of the study is to develop data that can convincingly guide clinicians on the use and efficacy of vedolizumab in patients with small bowel CD. There is an unmet need to identify response to vedolizumab in small bowel CD using objective endpoints. Current data suggest that MR enterography may meet this unmet need. There is an additional unmet need to develop predictive models incorporating both clinical and baseline radiological and endoscopic variables with higher discriminatory performance in identifying longer term clinical remission with vedolizumab. Finally, this proposal is strengthened by the exploratory studies which may identify new proteomic biomarkers that correlate with longer term radiological response with vedolizumab reflecting its latency of response. If successful, these serum biomarkers may guide a personalized approach to the treatment of small bowel CD with vedolizumab, allowing early identification of PNR, monitoring disease activity and the pharmacodynamics of vedolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe disease activity small bowel CD (small bowel only or ileocecal only) visible on MRE
* Initiated on Vedolizumab with/without thiopurines or methotrexate
* ≥18 years old

Exclusion Criteria:

* Pregnancy
* Age <18
* Planned surgery prior to the first follow-up MRE
* Inability to provide informed consent.
* Perianal CD will be excluded since assessment requires performance of additional MRI of the pelvis.
* Individuals with colonic involvement other than involvement of the ascending colon and cecum.
* Inpatient scans will only be included if this is a MRE and adequate small bowel distension with appropriate contrast has been achieved
* If unable to provide informed consent
* Contraindications for MRE including chronic kidney disease that precludes contrast administration, implanted medical devices that are contraindicated for MRE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parakkal Deepak, MBBS, MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deepak P, Fletcher JG, Fidler JL, Barlow JM, Sheedy SP, Kolbe AB, Harmsen WS, Loftus EV, Hansel SL, Becker BD, Bruining DH. Radiological Response Is Associated With Better Long-Term Outcomes and Is a Potential Treatment Target in Patients With Small Bowel Crohn's Disease. Am J Gastroenterol. 2016 Jul;111(7):997-1006. doi: 10.1038/ajg.2016.177. Epub 2016 May 10. PMID 27166131

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vedolizumab 300 MG Injection [Entyvio]
Started | 48
Week 14 Dose Escalation to Every 4 Weeks | 2
Completed | 22
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Vedolizumab 300 MG Injection [Entyvio]
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.95 [27.45 to 47.22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 7
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 48
Montreal Location [Number; unit: participants] — Montreal location classification for were disease is present
  participants
    L1 - terminal ileum | 8
    L3 - ileocolonic | 40
Montreal Behavior [Count of Participants; unit: Participants]
  B1 non-stricturing, non-penetrating | 22
  B1p non-stricturing, non-penetrating with perianal disease | 3
  B2 stricturing | 8
  B2p stricturing with perianal disease | 1
  B3 penetrating | 7
  B3p penetrating with perianal disease | 7
Montreal Age Classification [Count of Participants; unit: Participants]
  1 - Age of diagnosis at 16 years or younger | 6
  2 - Age of diagnosis at 17-40 years | 32
  3 - Age of diagnosis at >40 years | 10
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index (BMI) is a medical screening tool that measures the ratio of your height to your weight to estimate the amount of body fat you have. Healthcare providers calculate BMI by using weight in kilograms (kg) divided by the square of height in meters (m2).
  kg/m^2 | 28.10 [23.70 to 32.10]
Upper GI Involvement [Count of Participants; unit: Participants]
  No | 37
  Yes | 11
Perianal Involvement [Count of Participants; unit: Participants]
  No | 37
  Perianal Involvement | 11
Baseline Harvey Bradshaw Index Score [Mean (Inter-Quartile Range); unit: units on a scale] — The Harvey-Bradshaw Index (HBI) allow physicians to quickly categorize the severity of CD and detect remission. The total HBI score ranges from a minimum of "0" to "no theoretical maximum score." The theoretical maximum score is dependent on the number of liquid stools reported by the patient per day. A reported total HBI score of less than 5 indicates remission, 5-7 suggests mild severity, 8-16 denotes moderate severity, and greater than or equal to 16 demarks severe disease.
  units on a scale | 5 [2 to 9]
Baseline Crohn's Disease Activity Index Score [Mean (Inter-Quartile Range); unit: units on a scale] — The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from minimum of 0 to maximum of 600, with higher scores indicating greater disease activity. Clinical remission is defined by a CDAI score of ≤ 150 points.
  units on a scale | 143.00 [84.00 to 286.00]
Baseline EQ-5D Base_Mobility [Count of Participants; unit: Participants] — The descriptive system comprises the same 5 dimensions as the EQ5D-3L (mobility, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The reported values are the breakdown of how many participants responded to each level at Baseline.
  Participants
    1 - No problem walking | 36
    2 - Slight problems walking | 2
    3 - Moderate problems walking | 3
    4 - Severe problems walking | 0
    5 - Unable to walk | 0
    NA | 7
Baseline EQ-5D Base_Self-Care [Count of Participants; unit: Participants] — The descriptive system comprises the same 5 dimensions as the EQ5D-3L (mobility, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A total score is derived based on responses. The reported values are the breakdown of how many participants responded to each level at Baseline.
  Participants
    1 - No problems washing or dressing | 37
    2 - Slight problems washing or dressing | 3
    3 - Moderate problems washing or dressing | 1
    4 - Severe problems washing or dressing | 0
    5 - Unable to wash or dress | 0
    NA | 7
Baselin eEQ-5D Base_Usual Activities [Count of Participants; unit: Participants] — The descriptive system comprises the same 5 dimensions as the EQ5D-3L (mobility, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The reported values are the breakdown of how many participants responded to each level at Baseline.
  Participants
    1 - No problems doing usual activities | 26
    2 - Slight problems doing usual activities | 7
    3 - Moderate problems doing usual activities | 7
    4 - Severe problems doing usual activities | 1
    5 - Unable to do usual activities | 0
    NA | 7
Baseline EQ-5D Base_Pain Discomfort [Count of Participants; unit: Participants] — The descriptive system comprises the same 5 dimensions as the EQ5D-3L (mobility, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The reported values are the breakdown of how many participants responded to each level at Baseline.
  Participants
    1 - No pain or discomfort | 15
    2 - Slight pain or discomfort | 8
    3 - Moderate pain or discomfort | 10
    4 - Severe pain or discomfort | 6
    5 - Extreme pain or discomfort | 2
    NA | 7
Baseline EQ-5D Base_Anxiety [Count of Participants; unit: Participants] — The descriptive system comprises the same 5 dimensions as the EQ5D-3L (mobility, self care, usual activities, pain/discomfort, anxiety/depression). However, each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The reported values are the breakdown of how many participants responded to each level at Baseline.
  Participants
    1 - Not anxious or depressed | 22
    2 - Slightly anxious or depressed | 6
    3 - Moderately anxious or depressed | 6
    4 - Severely anxious or depressed | 7
    5 - Extremely anxious or depressed | 0
    NA | 7
Baseline EQ-5D Base_Your Health Today, 0-100 [Median (Inter-Quartile Range); unit: units on a scale of 0-100] — The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The EQ VAS has a scale of 0-100. This information can be used as a quantitative measure of health as judged by the individual respondents. The reported value is the median EQ-VAS score reported by all patients with a range of 65-90.
  units on a scale of 0-100 | 80 [65 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Radiological Response
Description: Radiological Transmural Response will be defined per-lesion and per-patient. Per-lesion TR will be defined as a decrease in the length of inflamed small bowel lesion from baseline or improvement in any imaging findings associated with severe mural inflammation, i.e., restricted diffusion, mural thickness, intramural T2 hyperintensity, peri-enteric T2 signal, and luminal ulcerations, without development of a new penetrating or stricturing complication. Worsened lesions will be fined as those with an increased score of any imaging parameter associated with severe mural inflammation. Unchanged lesions will be defined as those with unchanged (without worsening or improving) inflammatory parameters associated with severe mural inflammation. Patients will be then classified for TR as responders if all individual lesions improved and non-responders if any of the lesions worsened, a new lesion developed at the 4 month MRE and all other scenarios not meeting definition of response.
Time Frame: 24±2 weeks
Measure: Number; unit: participants
Arm/Group | Vedolizumab 300 MG Injection [Entyvio]
Number analyzed (Participants) | 22
participants
  Transmural Ulcer Healing | 21
  Transmural Remission | 16

2. Primary Outcome: Radiological Response
Description: as for outcome 1
Time Frame: 52±2 weeks
Measure: Number; unit: participants
Arm/Group | Vedolizumab 300 MG Injection [Entyvio]
Number analyzed (Participants) | 12
participants
  Transmural Ulcer Healing | 12
  Transmural Remission | 9

ADVERSE EVENTS:
Time Frame: Over the course of the participants time in the study, which was 1 year.
Groups:
- Vedolizumab 300 MG Injection [Entyvio] Every 8 Weeks; Vedolizumab 300 MG Injection [Entyvio] Every 4 Weeks (Dose Escalation) After Week 14: Vedolizumab will be initiated at 300 mg intravenous (IV) dosing at 0, 2 and 6 weeks followed by the 1st maintenance with 300 mg IV at week 14. Patients who have not achieved clinical response at week 14 will be eligible to undergo dose escalation to 4 weekly dosing of vedolizumab depending on the judgement of the treating gastroenterologist.
  Vedolizumab 300 MG Injection [Entyvio]: Vedolizumab Injection
Arm/Group | Vedolizumab 300 MG Injection [Entyvio] Every 8 Weeks | Vedolizumab 300 MG Injection [Entyvio] Every 4 Weeks (Dose Escalation) After Week 14
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/2
Other Adverse Events (participants affected / at risk) | 0/46 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03142321/Prot_SAP_001.pdf